CLINICAL TRIAL: NCT02672995
Title: Fractionated Stereotactic Radiosurgery With Concurrent Bevacizumab for Brain Metastases: A Phase I Dose-escalation Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201511005MINB
Record Dates: First submitted 2016-01-28; First posted 2016-02-03 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Brain Neoplasm
Keywords: stereotactic radiosurgery,Bevacizumab
MeSH Terms: conditions — Brain Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm dose-escalation (Experimental): Fractionated stereotactic radiosurgery:
  Group 1: tumors 1.5~2.5 cm in diameter Dose level 1: 21 Gy in 3 fractions Dose level 2: 24 Gy in 3 fractions Dose level 3: 27 Gy in 3 fractions Group 2: tumors 2.5~3.5 cm in diameter Dose level 1: 18 Gy in 3 fractions Dose level 2: 21 Gy in 3 fractions Dose level 3: 24 Gy in 3 fractions Three fractions will be given in one week with at least 1 day break.
  Concurrent bevacizumab:
  Bevacizumab 7.5 mg/kg will be given one day before the first fraction of radiosurgery and 2 weeks after the first dose of bevacizumab.
  Interventions: Radiation: Fractionated stereotactic radiosurgery; Drug: bevacizumab

INTERVENTIONS:
Radiation: Fractionated stereotactic radiosurgery — Fractionated stereotactic radiosurgery:
  Group 1: tumors 1.5~2.5 cm in diameter Dose level 1: 21 Gy in 3 fractions Dose level 2: 24 Gy in 3 fractions Dose level 3: 27 Gy in 3 fractions Group 2: tumors 2.5~3.5 cm in diameter Dose level 1: 18 Gy in 3 fractions Dose level 2: 21 Gy in 3 fractions Dose level 3: 24 Gy in 3 fractions Three fractions will be given in one week with at least 1 day break.
  Other Names: Fractionated SRS
Drug: bevacizumab — Concurrent bevacizumab:
  Bevacizumab 7.5 mg/kg will be given one day before the first fraction of radiosurgery and 2 weeks after the first dose of bevacizumab.
  Other Names: Avastin

SUMMARY:
The investigators propose a new treatment strategy of fractionated stereotactic radiosurgery with concurrent bevacizumab for brain metastases. This phase I dose-escalation study is to establish the feasibility of this strategy and find the recommended doses.

DETAILED DESCRIPTION:
For each group (two groups according to tumor size), the design proceeds with cohorts of three patients, with the first cohort treated at a starting dose. If none of the three patients in a cohort experiences a dose-limiting toxicity (DLT), the next cohort with three patients will be treated at the next higher dose level. If one of the first three patients experiences a dose-limiting toxicity, the next cohort will be treated at the same dose level. The dose escalation continues until at least two patients among a cohort of three to six patients experience DLTs and the maximum tolerated dose (MTD) will be the dose level just below. If the highest planned dose was achieved without two patients experiencing DLTs, the MTD will be that dose level.

The DLT is defined as grade 4 or above toxicities according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 within 4 months after stereotactic radiosurgery (SRS):

Grade 4 central nervous system necrosis (life-threatening consequences; urgent intervention indicated) Grade 4 sensory or motor neuropathy (life-threatening consequences; urgent intervention indicated) Grade 4 hemorrhage (life-threatening consequences; urgent intervention indicated) or Grade 4 thromboembolic event (life-threatening consequences such as pulmonary embolism, cerebrovascular event, arterial insufficiency; hemodynamic or neurologic instability; urgent intervention indicated) Grade 4 hypertension (life-threatening consequences such as malignant hypertension, transient or permanent neurologic deficit, hypertensive crisis; urgent intervention indicated)

Study treatment:

Fractionated stereotactic radiosurgery:

Group 1: tumors 1.5~2.5 cm in diameter Dose level 1: 21 Gy in 3 fractions Dose level 2: 24 Gy in 3 fractions Dose level 3: 27 Gy in 3 fractions Group 2: tumors 2.5~3.5 cm in diameter Dose level 1: 18 Gy in 3 fractions Dose level 2: 21 Gy in 3 fractions Dose level 3: 24 Gy in 3 fractions Three fractions will be given in one week with at least 1 day break.

Concurrent bevacizumab:

Bevacizumab 7.5 mg/kg will be given one day before the first fraction of radiosurgery and 2 weeks after the first dose of bevacizumab.

ELIGIBILITY:
Inclusion criteria

To be eligible for inclusion, patients must fulfill the following criteria:

1. Patients with a histologic diagnosis of non-hematopoietic malignancy and radiographic evidence of measurable brain metastases (1.5~3.5 cm).
2. The number of brain metastases receiving fractionated SRS: ≤3.
3. No evidence of leptomeningeal metastasis on gadolinium-enhanced MRI within 30 days prior registration.
4. Age ≥ 20 years.
5. Karnofsky Performance Status ≥ 60.
6. Life expectancy of ≥ 4 months.
7. Women of childbearing potential and male participants must practice adequate contraception.
8. Patients must be able to comply with the study protocol and follow-up schedules and provide study-specific informed consent.

Exclusion criteria Patients fulfill any of the following criteria will be excluded from this trial

1. Serum creatinine > 2.0 mg/dL within 30 days prior registration
2. Contraindication to magnetic resonance (MR) imaging such as implanted metal devices or foreign bodies, severe claustrophobia
3. Patients with evidence of bleeding diathesis or coagulopathy, international normalized ratio (INR) >1.5
4. Patients who require the use of warfarin sodium > 1 mg
5. Patients with active GI ulcers, GI bleeding, or active inflammatory bowel disease
6. Patients with clinically significant cardiac disease (e.g., uncontrolled hypertension [blood pressure of >160/90 mmHg on medication], history of myocardial infarction or unstable angina within 12 months of registration), New York Heart Association (NYHA) Class II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia) are not eligible
7. Patients with a history of aneurysms, cerebrovascular accident (CVA) and arteriovenous malformations
8. Patients with arterial thromboembolic events, including transient ischemic attack (TIA), or clinically significant peripheral artery disease within 6 months of registration
9. Patients with serious, non-healing wound, ulcer, or current healing fracture
10. Patients with a history of any type of fistula (vesicovaginal, gastrointestinal, etc) or gastrointestinal perforation
11. Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements, defined as follows:

    1. Uncontrolled active infection requiring intravenous antibiotics at the time of registration
    2. Transmural myocardial infarction ≤ 6 months prior to registration
    3. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
    4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
    5. Uncontrolled psychiatric disorder
12. Will receive any other investigational agent or chemotherapy and/or target therapies during SRS
13. Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 4 months
  The maximum tolerated dose of fractionated stereotactic radiosurgery with concurrent bevacizumab for brain metastases.

SECONDARY OUTCOMES:
Response rate | 4 months
  Response rate
Time to progression | 4 months
  Time to progression
The incidence of radiation-induced adverse effects | 4 months
  The incidence of radiation-induced adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chun Wang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided